CLINICAL TRIAL: NCT01928901
Title: Randomized, Placebo-controlled, Double-blind, Cross-over Trial With Bronchipret and Sinupret to Evaluate Acceleration of Mucociliary Clearance (MCC)
Brief Title: Trial With Bronchipret and Sinupret to Evaluate Acceleration of Mucociliary Clearance (MCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Saccharin test
Record Dates: First submitted 2013-08-14; First posted 2013-08-27 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Current Smokers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- administration of Bronchipret (Experimental): 7 days of administration of Bronchipret, 2 FCT t.i.d
  Interventions: Drug: administration of Bronchipret; Drug: administration of Bronchipret Placebo
- administration of Sinupret (Experimental): 7 days of administration of Sinupret, 2 CT t.i.d
  Interventions: Drug: administration of Sinupret; Drug: administration of Sinupret Placebo
- administration of Bronchipret Placebo (Placebo Comparator): 7 days of administration of Bronchipret Placebo, 2 FCT t.i.d
  Interventions: Drug: administration of Bronchipret; Drug: administration of Bronchipret Placebo
- administration of Sinupret Placebo (Placebo Comparator): 7 days of administration of Sinupret Placebo, 2 CT t.i.d
  Interventions: Drug: administration of Sinupret; Drug: administration of Sinupret Placebo

INTERVENTIONS:
Drug: administration of Sinupret
  Arms: administration of Sinupret; administration of Sinupret Placebo
Drug: administration of Bronchipret
  Arms: administration of Bronchipret; administration of Bronchipret Placebo
Drug: administration of Sinupret Placebo
  Arms: administration of Sinupret; administration of Sinupret Placebo
Drug: administration of Bronchipret Placebo
  Arms: administration of Bronchipret; administration of Bronchipret Placebo

SUMMARY:
Proof of concept: Superiority of Bronchipret or Sinupret to placebo in respect to mucociliary clearance

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers who have given their signed declaration of consent and have signed the data protection declaration
2. Male or female volunteers 25 - 40 years
3. Current smokers (5-20 cigarettes per day since 5 years at least)
4. Ability to taste sweetness of saccharin
5. Perception of sweetness within 30 minutes after placement of saccharin behind nasal valve

Exclusion Criteria:

1. Ciliary dyskinesia
2. Cystic fibrosis
3. COPD/emphysema
4. Asthma
5. Chronic rhinosinusitis
6. Acute respiratory tract infection within the last 6 weeks prior to enrolment
7. Septal or sinus surgery
8. Symptomatic allergic rhinitis
9. Known allergic rhinitis
10. Treatment with not-permitted previous or concomitant therapy
11. History of snuff consumption for longer than 1 month or intranasal consumption of recreational drugs such as cocaine or heroin for longer than 1 month
12. Any disease or condition that might affect the safety of the subject during the trial, according to the investigator's judgement

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Time to perception of sweetness | after 7 days of treatment
  Time to perception of sweetness after 7 days of treatment with the investigational products - relative to the time to perception of sweetness at the begin-ning of treatment

SECONDARY OUTCOMES:
Perception of Sweetness of Saccharin | 4 - 7 weeks
  To measure the time to perception of sweetness of Saccharin after 7 days of treatment with the investigational products calculated as difference to time to perception of sweetness at the beginning of treatment. The time of sweetness will be measured in minutes and seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, Prof.Dr.Dr., Study Chair — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Ghent, Belgium